CLINICAL TRIAL: NCT07322887
Title: A Phase 2, Randomized, Double-blind, Placebo-Controlled, Single-Center Study to Assess the Effects of SUL-238 on High Energy Phosphates With Magnetic Resonance Spectroscopy (³¹P-MRS) in Patients With Early, Untreated Parkinson's Disease ("SHEPHERD" STUDY)
Brief Title: A Phase 2 Study to Assess the Effects of SUL-238 on High Energy Phosphates With ³¹P-MRS in Patients With Early, Untreated Parkinson's Disease
Acronym: SHEPHERD
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: GEN İlaç ve Sağlık Ürünleri A.Ş. (Industry)
Collaborators: Sulfateq B.V. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GN-002; 2025-524674-42-00 (EU CTIS Number)
Record Dates: First submitted 2025-11-28; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Parkinson's Disease (PD)
Keywords: Phase 2; SUL-238; Mitochondrial function; Magnetic Resonance Spectroscopy; MRS
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SUL-238 high dose (Experimental): SUL-238 (1500 mg t.i.d.)
  Interventions: Drug: SUL-238 (1500 mg t.i.d.) film-coated tablets
- SUL-238 low dose (Experimental): SUL-238 (500 mg t.i.d.)
  Interventions: Drug: SUL-238 (500 mg t.i.d.) film-coated tablets
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SUL-238 (1500 mg t.i.d.) film-coated tablets — Oral treatment with high dose SUL-238 for 28 days
  Arms: SUL-238 high dose
Drug: SUL-238 (500 mg t.i.d.) film-coated tablets — Oral treatment with low dose SUL-238 for 28 days
  Arms: SUL-238 low dose
Drug: Placebo — Oral treatment with placebo for 28 days
  Arms: Placebo

SUMMARY:
The main goal of the study is to investigate how well the new drug SUL-238 works in Parkinson's Disease (PD). This is done by means of an MRS scan. An MRS scan is similar to a regular MRI scan. It will also learn about the safety of new drug SUL-238. The main questions it aims to answer are:

* Does new drug SUL-238 improve the mitochondrial function in patients with Parkinson's Disease (PD)?
* What medical problems do participants have when taking new drug SUL-238?

Researchers will compare new drug SUL-238 to a placebo (a look-alike substance that contains no drug) to see if SUL-238 works to improve mitochondrial function in patients with PD.

Participants will:

* Take new drug SUL-238 or a placebo every day for 28 days
* Visit the clinic once every 2 weeks for checkups and tests during the treatment period and finally 28 days after the last dose of SUL-238
* Keep a diary of their symptoms and the number of times they use oral new drug SUL-238

DETAILED DESCRIPTION:
Two different oral doses of SUL-238 (1500 mg t.i.d. or 500 mg t.i.d) or placebo will be administered to patients with early, untreated Parkinson's Disease (PD), aged ≥40 years. Patients will be randomly assigned to one of the 3 groups using 1:1:1 randomization, each group will consist of 15 patients. Patients will be stratified based on their sex in to ensure similar distribution of both sexes in each group. Drop-outs will be replaced with new patients to reach 15 patients in each group. Study drugs will be administered after fasting from all food and drink except water for a minimum of 1 hour prior to dosing. Patients will be allowed to eat 1 hour after receiving their dose. Only morning dose will be given on day 28, there will be no dosing between day 29 and 56.

There will be three study periods per treatment group:

* A maximum of four-week screening period (Screening Period)
* A four-week treatment period (Treatment Period)
* A four-week follow-up period (End-of-Study Assessment)

Patients will be visiting the study center in the morning, in total five times for study assessments and collections of blood samples until day 56. Blood samples will be collected on days 1, 14, 28, and 56 (On day 1 [pre-dose baseline, post-dose at 1 hr], and days 14 [pre-dose], 28 [post-morning dose at 1 hr and 4 hr]).

Patients who agreed to provide CSF in each group will give one CSF sample on day 28 at 4 hours post-morning dose.

Voxel Metabolite Measurements:

MRI/MRS scans will be conducted on a Siemens 3 MAGNETOM Cima.X scanner located at the at the UMCG. Patients will undergo 31P-MRS scans to measure concentrations of the following mitochondria-related brain metabolites: ATP, phosphocreatine and inorganic phosphate, as well as membrane related phospholipids PME and PDE.

Preparation: A 31P/1H T/R head coil will be used. The head of the patient will be positioned at the center of the coil. Prior to 31P-MRS, T1 and T2 weighted structural images are acquired for reference purposes during voxel placement.

31P-MRS scans: 31P spectra will be acquired from voxels placed in the precentral gyrus, substantia nigra and putamen regions (each contralateral to the most affected side of the body). Spectra for the precentral gyrus and putamen will be recorded at rest, during fist clenching on the contralateral side and during recovery. For substantia nigra, spectra will only be acquired during rest. For each ROI the total acquisition will be at most 15 minutes.

ELIGIBILITY:
Inclusion Criteria:

1. Untreated Parkinson's Disease (PD) patients diagnosed in accordance with the UK PDS Brain Bank Criteria for the diagnosis of PD. Patients must have bradykinesia and at least one of the following:

   1. muscular rigidity
   2. rest tremor (4-6 Hz)
   3. postural instability unrelated to primary visual, cerebellar, vestibular or proprioceptive dysfunction.
2. The duration of PD since diagnosis is ≤ 1 year.
3. Patients with Modified Hoehn and Yahr stage ≤ 1.0.
4. Patients with Montreal Cognitive Assessment (MOCA) score of ≥22.
5. Men and women aged ≥40 years at screening.
6. Able to understand the nature of the study and provide signed and dated written informed consent in accordance with local regulations before the conduct of any study related procedures.
7. Able to complete all study related testing and evaluations.
8. Patients must be, in the opinion of the Investigator, able to participate in all scheduled evaluations, likely to complete all required tests, and likely to be compliant.
9. Men and women of child-bearing potential with partners of child-bearing potential must agree to use highly effective contraception. For male and female patients, contraception should continue for 90 days after the last dose of investigational medicinal product (IMP, one spermatic cycle).
10. Women of non-childbearing potential must be post-menopausal (the last menstrual period was at least 12 months ago, and follicle-stimulating hormone [FSH] at screening confirms post-menopausal status), or have no uterus, ovaries, or fallopian tubes (or have their fallopian tubes tied). All women must have a negative pregnancy test result before administration of test article. Women who are surgically sterile must provide documentation of the procedure by an operative report or by ultrasound.

Exclusion Criteria:

1. Atypical parkinsonism, including that due to drugs, metabolic disorders, encephalitis, cerebrovascular disease, normal pressure hydrocephalus, or other neurodegenerative disease.
2. Any history of intellectual disability or psychiatric disorders, including substance use disorders, according to the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) criteria, except a history of mild depression/anxiety that has been resolved for at least the past 3 months.
3. A positive Hepatitis B surface antigen, Hepatitis C antibody, or Human Immunodeficiency Virus (HIV) antibody test at screening.
4. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) levels greater than 1.5 times the upper limit of normal (ULN) at screening or between screening and first dose administration.
5. Received or used an investigational product (including placebo) or device within the following time period prior to day -1 in the current study: 90 days, 5 half-lives, or twice the duration of the biological effect of the investigational product (whichever is longer).
6. Use of non-prescription drugs, vitamins, herbal, and dietary supplements which has potential to influence the mitochondrial function (such as coenzyme Q10, carnitine, creatine, lipoic acid and vitamin E) within 30 days prior to day -1.
7. History of clinically significant sensitivity to any of the study medications, or components thereof or a history of drug or other allergies that, in the opinion of the Investigator or Medical Monitor, contraindicates their participation.
8. Women with a positive pregnancy test, are lactating, or are planning to become pregnant during the study or within 6 months of the end of this study.
9. A history or presence of any disease, condition, or surgery likely to affect drug absorption, distribution, metabolism, or excretion. Patients with a history of cholecystectomy should be excluded.
10. A history or presence of a clinically significant hepatic, renal, gastrointestinal, cardiovascular, endocrine, pulmonary, ophthalmologic, immunologic, hematologic, dermatologic, or neurologic (other than PD) abnormality.
11. At screening, any clinically significant abnormalities in rhythm, conduction, or morphology of the resting ECG and any abnormalities in the 12-lead ECG that, in the judgement of the Investigator or Medical Monitor, may interfere with the interpretation of QTc interval changes, including abnormal ST-T-wave morphology or left ventricular hypertrophy.
12. A clinically significant vital signs abnormality at screening or day -1. This includes, but is not limited to, the following, in the sitting position (3 measurements, each 5 minutes apart):

    1. systolic blood pressure (SBP) < 90 or >140 mmHg,
    2. diastolic blood pressure (DBP) < 50 or > 95 mmHg, or
    3. heart rate < 45 or > 100 beats per minute.
13. In the opinion of the Investigator or Medical Monitor, the patient is unlikely to comply with the protocol or is unsuitable for any reason, e.g., known issues with ability to swallow tablets.
14. Women of child-bearing potential, or men, who are unwilling or unable to use accepted methods of birth control for up to 3 months following study participation.
15. Contraindications for undergoing an MRI.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2026-03-02 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Assessment of the effect of SUL-238 on mitochondria-related brain metabolites in Parkinson's Disease (PD) Patients | At baseline and end of treatment at 4 weeks
  Mean change from baseline to Week 4 in each active dose group as compared to placebo in the concentration of mitochondria-related brain metabolites (ATP, phosphocreatine and inorganic phosphate), as measured by ³¹P-Magnetic Resonance Spectroscopic (MRS) imaging, in the following regions of interest: 1. Putamen, 2. Substantia Nigra, 3. Motor Cortex

SECONDARY OUTCOMES:
Assessment of the effect of SUL-238 treatment on systemic biomarkers of mitochondrial function and associated pathways in Parkinson's Disease (PD) patients by predefined mitochondria related plasma targeted metabolomics | At baseline and end of treatment at 4 weeks
  Mean change from baseline to Week 4 in each active dose group as compared to placebo in the circulating levels of established indicators of mitochondrial dysfunction such as lactate, pyruvate and lysophosphatidylcholine
Assessment of the effect of SUL-238 treatment on systemic biomarkers of mitochondrial function and associated pathways in Parkinson's Disease (PD) patients by predefined mitochondria related plasma targeted proteomics | At baseline and end of treatment at 4 weeks
  Mean change from baseline to Week 4 in each active dose group as compared to placebo in the circulating levels of established indicators of mitochondrial dysfunction such as cell-free Cytochrome c, creatinine and succinate dehydrogenase (SDH)
Assessment of safety and tolerability of SUL-238 in Parkinson's Disease (PD) Patients | From enrollment to the end of follow-up period at 8 weeks
  Safety and tolerability of SUL-238 will be assessed by the number of participants;
  1. with adverse events,
  2. with abnormal laboratory test results,
  3. abnormal vital signs,
  4. abnormal electrocardiogram,
  5. abnormal physical and neurological examination

OTHER OUTCOMES:
Assessment of the effect of SUL-238 compared to placebo in improving motor symptoms in Parkinson's Disease (PD) Patients | At baseline and end of treatment at 4 weeks
  Mean change from baseline to Week 4 in The Movement Disorder Society-Sponsored Revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part III (score range: 0-132, higher scores mean a worse outcome) compared with placebo
Assessment of the effect of SUL-238 compared to placebo on global cognitive function in Parkinson's Disease (PD) Patients | At baseline and end of treatment at 4 weeks
  Mean change from baseline to Week 4 in the Montreal Cognitive Assessment (MoCA) score (score range: 0-30, higher scores mean a better outcome), compared with placebo
Characterization of the plasma pharmacokinetic profile of SUL-238 | From enrollment to the end of follow-up treatment at 4 weeks
  Quantify SUL-238 (as SUL-138) concentrations in plasma at specified time points:
  1. Day 1: Pre-dose, 1-hour postdose
  2. Day 14: Pre-dose
  3. Day 28: Pre-dose, 1-hour postdose, 4-hours post-dose
Characterization of the pharmacokinetic profile of SUL-238 in cerebrospinal fluid (CSF) | At the end of treatment at week 4
  Quantify SUL-238 (as SUL-138) concentration in CSF at a single time point: 4-hours post-dose on Day 28 (in consenting patients).
Identification and assessment of potential pharmacodynamic effects of SUL-238 | From enrollment to the end of follow-up treatment at 4 weeks
  Mean changes from baseline in the levels of exploratory plasma biomarkers such as level of plasma cell-free mtDNA at Days 14 and 28

CONTACTS AND LOCATIONS:
Locations (1):
- CTC Netherlands BV, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No